CLINICAL TRIAL: NCT02414321
Title: The Role of the Pulmonary Vasculature in the Fontan Circulation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Prof. dr. R.M.F. Berger, Professor and Head of Department of Pediatric Cardiology, University Medical Center Groningen
Other Study IDs: NL51128.042.15
Record Dates: First submitted 2015-03-30; First posted 2015-04-10 (Estimated); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Congenital Heart Disease; Fontan Operation; Pulmonary Vascular Resistance; Pulmonary Vascular Remodeling
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Fontan group: Right heart catheterization:
  * pulmonary artery OCT analysis
  * dobutamine stress test
  * pulmonary vascular response test (nitric oxide)
  * trans-thoracic echocardiography
- Control group: Right heart catheterization:
  - pulmonary artery OCT analysis
- PAH group: Right heart catheterization:
  - pulmonary artery OCT analysis

SUMMARY:
This study aims to explore the structural and functional characteristics of the pulmonary vasculature in adult Fontan patients.

Objectives:

* Determine the effect of pulmonary vasodilatation on indexed cardiac output during simulated exercise.
* Characterization of structural properties of small pulmonary arteries.

DETAILED DESCRIPTION:
Rationale:

The Fontan circulation is a palliation for patients with a functionally univentricular heart. The Fontan circulation is characterized by impaired exercise capacity and gradual attrition over time. To date treatment options are extremely limited. It has been proposed that pulmonary vascular resistance (PVR) is the controlling and limiting factor of cardiac output in the Fontan circulation. Remodeling of the pulmonary vasculature and increasing PVR are possible key factors in the long term failure of the Fontan circulation. Optical Coherence Tomography (OCT) is an intravascular imaging modality used for structural characterization of blood vessels. Nitric oxide is a pulmonary vasodilator used in pulmonary vascular response tests, aimed at lowering PVR which may improve cardiac output in the Fontan circulation. These two diagnostic procedures are tools to study the structural and functional characteristics of the pulmonary vasculature in the Fontan circulation. The results of this study could identify the pulmonary circulation as a future treatment target in Fontan patients and may provide clues for new therapeutic treatment strategies to improve the long term outcome of these patients.

Study procedure:

The study protocol will be performed during a clinically indicated cardiac catheterization. In the context of this study additional measurements will be performed which will include a pulmonary vascular response test, trans-thoracic echocardiography and pulmonary artery OCT measurements.

ELIGIBILITY:
Inclusion criteria:

Fontan group

* written informed consent
* Clinical indication for cardiac catheterization

Control group

* written informed consent
* Clinical indication for right heart catheterization
* Absence of pulmonary vascular disease
* Normal pulmonary vascular hemodynamic profile

Exclusion criteria:

Fontan group

* Standard exclusion criteria for cardiac catheterization
* Obstruction in Fontan conduit
* Inability to measure a reliable cardiac index and PVR (rhythm instability, hemodynamic or anatomic reasons)

Control Group

- No specific exclusion criteria apart from the standard exclusion criteria for right heart catheterization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (≥18 years), who attend the University Medical Center Groningen for follow-up after a Fontan completion.
  Additionally 5 adult patients (≥18 years) without a Fontan circulation and without a univentricular heart-like diagnosis but with a clinical indication for right heart catheterization and normal values at right heart catheterization measurements will be included to serve as controls for the pulmonary artery OCT analysis.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-06; Primary Completion 2024-06-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
vasodilatation | change in indexed cardiac output between baseline and after 10 minutes of pulmonary vasodilatation at heart catheterization
  change in indexed cardiac output between baseline and after pulmonary vasodilatation
number of intimal lesions in small pulmonary arteries | baseline at heart catheterization
  number of intimal lesions in small pulmonary arteries

CONTACTS AND LOCATIONS:
Overall Officials: Rolf M Berger, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Background] Fontan F, Baudet E. Surgical repair of tricuspid atresia. Thorax. 1971 May;26(3):240-8. doi: 10.1136/thx.26.3.240. PMID 5089489
- [Background] Wolff D, van Melle JP, Ebels T, Hillege H, van Slooten YJ, Berger RM. Trends in mortality (1975-2011) after one- and two-stage Fontan surgery, including bidirectional Glenn through Fontan completion. Eur J Cardiothorac Surg. 2014 Apr;45(4):602-9. doi: 10.1093/ejcts/ezt461. Epub 2013 Sep 25. PMID 24067749
- [Background] de Leval MR, Deanfield JE. Four decades of Fontan palliation. Nat Rev Cardiol. 2010 Sep;7(9):520-7. doi: 10.1038/nrcardio.2010.99. Epub 2010 Jun 29. PMID 20585329
- [Background] Gewillig M, Brown SC, Eyskens B, Heying R, Ganame J, Budts W, La Gerche A, Gorenflo M. The Fontan circulation: who controls cardiac output? Interact Cardiovasc Thorac Surg. 2010 Mar;10(3):428-33. doi: 10.1510/icvts.2009.218594. Epub 2009 Dec 7. PMID 19995891
- [Background] Goldberg DJ, Avitabile CM, McBride MG, Paridon SM. Exercise capacity in the Fontan circulation. Cardiol Young. 2013 Dec;23(6):824-30. doi: 10.1017/S1047951113001649. PMID 24401254
- [Background] Khambadkone S, Li J, de Leval MR, Cullen S, Deanfield JE, Redington AN. Basal pulmonary vascular resistance and nitric oxide responsiveness late after Fontan-type operation. Circulation. 2003 Jul 1;107(25):3204-8. doi: 10.1161/01.CIR.0000074210.49434.40. Epub 2003 Jun 23. PMID 12821557
- [Background] Ridderbos FJ, Wolff D, Timmer A, van Melle JP, Ebels T, Dickinson MG, Timens W, Berger RM. Adverse pulmonary vascular remodeling in the Fontan circulation. J Heart Lung Transplant. 2015 Mar;34(3):404-13. doi: 10.1016/j.healun.2015.01.005. Epub 2015 Jan 16. PMID 25813767